CLINICAL TRIAL: NCT03656692
Title: A Multicenter, Open Label Pilot Study to Explore the Efficacy and Safety of Acthar Gel in Subjects With Severe Noninfectious Intermediate Uveitis, Posterior Uveitis, or Panuveitis (NIPPU)
Brief Title: Safety and Effectiveness of Acthar Gel for Inflammation of the Eye's Uvea (Middle Layer)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Logistical challenges; no safety concerns
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNK61074105
Record Dates: First submitted 2018-08-21; First posted 2018-09-04 (Actual); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Uveitis, Posterior; Uveitis, Intermediate; Panuveitis
MeSH Terms: conditions — Uveitis, Posterior; Uveitis, Intermediate; Panuveitis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Acthar Gel (Other): Participants received Acthar 1 mL (80 units [U]) subcutaneously (SC) 2 times per week for 36 weeks followed by a taper to Acthar 1 mL (80 U) SC once a week for 2 weeks, then 0.5 mL (40 U) SC once a week for 2 weeks.
  Interventions: Drug: Acthar Gel

INTERVENTIONS:
Drug: Acthar Gel — Acthar gel for subcutaneous injection 80 units per mL (40 units per 0.5 mL)
  Other Names: Corticotropin

SUMMARY:
The main reason for this study is to see if Acthar Gel can reduce inflammation in the uvea.

Also, safety information when using it for this purpose will be collected.

ELIGIBILITY:
Inclusion criteria:

* Is male or nonpregnant, nonlactating female
* Has been diagnosed with current severe NIPPU
* Has active disease at the Baseline Visit as defined by the presence of at least 1 of the following parameters in at least one eye despite at least 2 weeks of maintenance therapy with oral prednisone (or oral corticosteroid equivalent):

  1. Has active, inflammatory, chorioretinal and/or inflammatory retinal vascular lesion
  2. Has ≥ 2+ anterior chamber cells [Standardization of Uveitis Nomenclature (SUN) criteria]
  3. Has ≥ 1.5+ vitreous haze
* Is willing to taper current doses of corticosteroid and immunomodulatory therapy to the minimum effective dose during the study.
* If under treatment with any immunosuppressants, immunomodulators, or biologic agents for a comorbid condition, has been on a stable dose for 2 weeks before screening

Exclusion criteria:

* Has proliferative or severe nonproliferative diabetic retinopathy, clinically significant macular edema due to diabetic retinopathy, neovascular/wet age-related macular degeneration, abnormality of vitreoretinal interface with the potential for macular structural damage independent of the inflammatory process or severe vitreous haze that precludes visualization of the fundus at the Baseline Visit
* Has Type 1 or Type 2 diabetes mellitus, tuberculosis, history of hepatitis, peptic ulcer, active infection, or any contraindication for treatment with Acthar Gel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Lead, Study Director — Mallinckrodt
Locations (8):
- United States (8):
  - Blue Ocean Clinical Research, Clearwater, Florida
  - Midwest Eye Institute, Indianapolis, Indiana
  - Massachusetts Eye Research and Surgery Institution (MERSI), Waltham, Massachusetts
  - Metropolitan Eye Research and Surgery Institute, Palisades Park, New Jersey
  - Bergstrom Eye Research, LLC, Fargo, North Dakota
  - Valley Retina Institute, PA, McAllen, Texas
  - Foresight Studies, LLC, San Antonio, Texas
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No
Discussion of statistical endpoints and analysis are included in manuscripts. Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT03656692) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 30 participants were planned, but only 5 enrolled before the study was terminated
Groups:
- Acthar Gel: Participants receive Acthar Gel
Period: Overall Study
Arm/Group | Acthar Gel
Started | 5
Completed | 2
Not Completed | 3
Not completed — Worsening of disease activity | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat population included all participants who received at least one dose of study treatment.
Arm/Group | Acthar Gel
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 58.0 [30.0 to 61.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Score on the Nussenblatt Grading Scale
Description: The Nussenblatt grading scale uses photographic measurement of cloudy, declining vision (vitreous haze). The scale goes from 0 to 4, and lower scores are better.
Time Frame: Week 36
Population: Data were not collected.
Arm/Group | Acthar Gel
Number analyzed (Participants) | 0

2. Primary Outcome: Score on the Laser Flare Scale
Description: Protein that escapes from blood vessels inside the eye make a sudden burst of scattered light (flare) when a laser shines on them. This is called a laser flare. It is used to measure the amount and size of proteins in the clear fluid in the front of the eyeball (aqueous humour). The larger the flare, the more inflammation is inside the eye (intraocular inflammation) in patients with uveitis. Laser flare is scored on a scale from 0 (no visible flare when compared with the normal eye) to 3 (severe - very dense flare). Lower scores are better.
Time Frame: Week 36
Population: Data were not collected.
Arm/Group | Acthar Gel
Number analyzed (Participants) | 0

3. Primary Outcome: Score on the Aqueous Cell Scale
Description: The number of cells (like white blood cells) floating in the aqueous humour (aqueous cells) are measured on a scale from 0 (none) to 4 (more than 30 cells), and lower scores are better.
Time Frame: Week 36
Population: Data were not collected.
Arm/Group | Acthar Gel
Number analyzed (Participants) | 0

4. Secondary Outcome: Diurnal Intraocular Pressure (IOP)
Description: Eye pressure is measured in millimeters of mercury (mmHg). Normal eye pressure ranges from 12-22 mmHg, and eye pressure greater than 22 mmHg is considered higher than normal. During a 24-hour period, IOP normally varies by 2 to 6 mmHg because of different amounts of secretion and drainage at different times of the day. The word diurnal means "around the day," and IOP means "pressure inside the eye", so diurnal IOP is the measure of pressure inside the eye during a 24-hour period. Diurnal IOP is measured in millimeters of mercury (mmHg) using Goldmann Applanation Tonometry (GAT). Lower scores are better.
Time Frame: Week 36
Population: Data were not collected.
Arm/Group | Acthar Gel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 44 weeks
Description: Treatment Emergent non-serious adverse events and all serious adverse events are reported. Treatment emergent adverse events are those that started or got worse after the first dose of study drug. Clinically significant change in vital signs, laboratory values and/or physical examinations are recorded as adverse events.
Arm/Group | Acthar Gel
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acthar Gel (N=5)
Iris adhesions (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Intraocular pressure increased (Investigations) | 2
Insomnia (Psychiatric disorders) | 2
Uveitis (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT03656692/Prot_SAP_000.pdf